CLINICAL TRIAL: NCT06983158
Title: A Phase 1/2a, Open-Label, Multi-Center, Dose-Escalation Trial to Assess Safety, Tolerability, and Efficacy of a Single Dose of CAP-002 Gene Therapy Administered to Pediatric Patients With Syntaxin-Binding Protein 1 (STXBP1) Encephalopathy
Brief Title: A Clinical Trial of CAP-002 Gene Therapy in Pediatric Patients With Syntaxin-Binding Protein 1 (STXBP1) Encephalopathy
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Per protocol stopping rule was met. Comprehensive review is needed prior to resuming enrollment.
Sponsor: Capsida Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CAP-002-101; SYNRGY (Other: Capsida Biotherapeutics)
Record Dates: First submitted 2025-05-05; First posted 2025-05-21 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-07

CONDITIONS: Developmental and Epileptic Encephalopathy
Keywords: STXBP1; Gene therapy
MeSH Terms: interventions — Genetic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Level 1 (Experimental): Participants will receive a single dose of STXBP1, administered IV
  Interventions: Drug: gene therapy
- Dose Level 2 (Experimental): Participants will receive a single dose of STXBP1, administered IV
  Interventions: Drug: gene therapy

INTERVENTIONS:
Drug: gene therapy — Intra-venous gene therapy

SUMMARY:
The goal of this clinical trial is to learn about the safety of CAP-002 gene therapy in children with Syntaxin-Binding Protein 1 (STXBP1) Encephalopathy. It will also provide information about whether CAP-002 demonstrates efficacy in treating children with STXBP1 with and without seizures.

Participants will have a single infusion of CAP-002, visit the clinic regularly for 2 years for checkups and tests and have seizures recorded in a diary by their caregiver.

DETAILED DESCRIPTION:
This is a Phase 1/2a, FIH, open-label, multi-center, dose-escalation trial to assess the safety, tolerability, and efficacy of a single intravenous (IV) dose of CAP-002 administered to participants with syntaxin-binding protein#1 (STXBP1) encephalopathy ages ≥18 months to <8 years of age.

Approximately 12 participants will be dosed in this trial. Phase 1 is a dose escalation phase that will dose approximately 6 participants divided into 2 cohorts (Cohort 1 and Cohort 2) while Phase 2a will have 1 dose cohort and dose approximately 6 participants. Participants in Phase 1 will be dosed sequentially in each cohort. Phase 2a will allow participants to be dosed concurrently if safety and tolerability data from Phase 1 are deemed acceptable.

Participants will receive a single intravenous infusion of CAP-002 and will then be followed for 2 years with safety measures, assessments to measure changes from Baseline in development, language, cognition, motor skills and behavior, a seizure diary and structured caregiver interviews.

Upon completion of the study or at the participant's final visit they will be invited to participate in a 3 year safety follow up study.

ELIGIBILITY:
Inclusion Criteria:

Male or female, ≥18 months to <8 years of age;

Has diagnosis of developmental encephalopathy due to an STXBP1 mutation with confirmation of a pathogenic or likely pathogenic STXBP1 gene mutation.

Has a legally authorized representative (LAR) willing and able to complete the informed consent process, willing to comply with trial procedures, and able to travel for repeat visits.

Is stable on any medication regimens (if being administered to control the signs and symptoms of underlying disease) for at least 6 weeks prior to trial entry and expected to be stable for at least 12 weeks post-CAP-002 administration.

Exclusion Criteria:

History of prior gene therapy;

Treatment with antisense oligonucleotide therapy within 6 months;

Presence of a confirmed mutation in a gene other than STXBP1 that is known to contribute to a neurodevelopmental disability or epilepsy;

Has presence of a significant non-STXBP1-related central nervous impairment/behavioral disturbance that would confound the scientific rigor or interpretation of results of the trial;

History of prematurity (defined as gestational age <35 weeks), history of low birth weight (<2.5 kg) and/or intra-uterine growth restriction, significant interventricular hemorrhage, structural brain deficit, or congenital heart disease;

Known contraindication to immunosuppression or other protocol-defined medications, including but not limited to corticosteroids or PPIs;

Clinically significant abnormalities in safety lab tests, vital signs;

Other illnesses or medications that may affect the interpretation of the study results;

Positive anti-capsid antibody test result.

Ages: 18 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2028-12-20 (Estimated); Study Completion 2028-12-20 (Estimated)

PRIMARY OUTCOMES:
Primary Safety | 2 years
  Incidence of Adverse Events and Serious Adverse Events assessed through Clinical safety laboratory tests (hematology, chemistry, liver function, and urinalysis), ECG, vital sign measurements, and Physical Examinations

SECONDARY OUTCOMES:
Bayley Scales of Infant and Toddler Development- Fourth Edition | Baseline, Month 6, Month 12, Month 18 and Month 24
  Clinician Scores: 0 to 2; Total Scores: Cognitive 0-162; Receptive 0-84; Expressive 0-74; Fine Motor 0-92; Gross Motor 0-116; High score is a better outcome
Gross Motor Function Measure | Baseline, Month 6, Month 12, Month 18 and Month 24
  Clinician Scores: 0 to 3; Total Score: 0 to 264; High score is a better outcome
Peabody Developmental Motor Scales-Third Edition | Baseline, Month 6, Month 12, Month 18 and Month 24
  Clinician Scores: 0 to 2; High score is a better outcome
STXBP1-Clinical Severity Assessment-Clinician | Baseline, Month 6, Month 12, Month 18 and Month 24
  Clinician Scores: 0 to 100; High score is a worse outcome
Vineland Adaptive Behavior Scales | Third Edition | Baseline, Month 6, Month 12, Month 18 and Month 24
  Caregiver Scores: 0 to 2; Total Scores: Receptive 0-78; Expressive 0-98, Written 0-76, Personal 0-110, Domestic 0-60, Community 0-116, Interpersonal 0- 86, Play and Leisure 0-72, Coping 0-66, Fine Motor 0- 68; Gross Motor 0-86: High score is a better outcome
Observer-Reported Communication Ability | Baseline, Month 6, Month 12, Month 18 and Month 24
  Caregiver Scores: No or only once; Sometimes, Yes, almost all the time; Yes, almost all the time is better outcome
Sensory Profile-2 | Baseline, Month 6, Month 12, Month 18 and Month 24
  Caregiver Scores: 1 to 5; Total Score: 0 to 625; High score is a worse outcome
Quality of Life Inventory-Disability | Baseline, Week 6, Month 6, Month 12, Month 18 and Month 24
  Caregiver Scores: Never, Rarely, Sometimes, Often, Very often; Very Often is better outcome
STXBP1-Clinical Severity Assessment-Caregiver | Baseline, Week 4, Week 8, Week 12, Month 4, Month 6, Month 12, Month 18 and Month 24
  Caregiver Scores: 0 to 100; High score is a worse outcome
Aberrant Behavior Checklist | Baseline, Month 6, Month 12, Month 18 and Month 24
  Caregiver Scores: 0 to 3; Total Score: 0-174; High score is a worse outcome
Child Behavior Checklist | Baseline, Month 6, Month 12, Month 18 and Month 24
  Caregiver Scores: 0 to 2; Total Behavior: 0 to 224; High score is a worse outcome
Child's Sleep Habits | Baseline, Month 6, Month 12, Month 18 and Month 24
  Caregiver Scores: 1 to 3; High score is a worse outcome
Seizure frequency | Baseline and daily though Month 24
  Caregiver assessment: Change from baseline in seizure experience as recorded in a seizure diary

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Brandabur, MD, Study Director — Capsida Biotherapeutics
Locations (4):
- United States (4):
  - Colorado Child Health Research Institute, Aurora, Colorado
  - Weill Cornell Medicine, New York, New York
  - Buerger Center for Advanced Pediatric Care, Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No